CLINICAL TRIAL: NCT03013374
Title: Protein Balance and Body Composition in Preterm Infants According to Feeding Regimen
Brief Title: Protein Balance and Body Composition in Preterm Infants
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Sponsor
Other Study IDs: Protein balance and FFM
Record Dates: First submitted 2016-12-30; First posted 2017-01-06 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2017-01

CONDITIONS: PreTerm Birth; Human Milk
Keywords: protein accretion; body composition
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Human milk fed infants: Infants fed fortified human milk at enrollment
  Any intervention is performed. Groups distinction is made according to own mother's milk availability.
- Preterm formula: Infants fed preterm formula milk at enrollment.
  Any intervention is performed. Groups distinction is made according to own mother's milk availability.

SUMMARY:
The adequacy of the quality of protein supply could influence the rate and the relative composition of weight gain in very low birth weight preterm infants.

Aim of the study is to investigate protein balance according to feeding regimen and the association between human milk feeding and fat free mass content at term corrected age in a cohort of very low birth weight infants.

DETAILED DESCRIPTION:
Nutritional management of preterm infants aims to approximate tissue growth and body composition of a foetus of same postconceptional age. The adequacy of the quality of protein supply could influence the rate and the relative composition of weight gain.

Aim of the study is to investigate protein balance according to feeding regimen and the association between exclusive human milk feeding and fat free mass content at term corrected age in a cohort of very low birth weight infants.

A prospective observational study. Infants are included according to inclusion criteria. Enrollment is performed at hospital discharge. Infants are divided into two groups (exclusively human milk or exclusively formula) according to own mother's milk availability. At enrollment macronutrients' intakes and protein balance are determined. Anthropometric measurements and body composition are also assessed. Nutritional composition of human milk is calculated by infrared spectroscopy (MIRIS® AB, Uppsala, Sweden). Protein balance is determined according to nitrogen balance standard method. Body composition is assessed by an air-displacement plethysmography system system (PEA POD Infant Body Composition System, COSMED SRL, Roma, Italy). At term corrected age anthropometry and body composition assessments are repeated.

ELIGIBILITY:
Inclusion Criteria:

* gestational age ≤32 weeks
* birth weight < 1500 grams
* birth weight ≥10th percentile according to Fenton's growth chart
* stable clinical conditions at discharge
* feeding by mouth with either exclusively human milk or formula at discharge

Exclusion Criteria:

* congenital or chromosomal abnormalities
* conditions that could interfere with growth such as chronic lung disease, neurological disorders, metabolic, cardiac disease and abdominal surgery, renal failure and/or sepsis (defined as a positive blood culture).

Ages: 23 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants are enrolled at time of hospital discharge. Infants with gestational age ≤32 weeks, birth weight < 1500 grams and ≥10th percentile according to Fenton's growth chart, having stable clinical conditions and feeding by mouth with either exclusively human milk or formula at discharge were included. Exclusion criteria were the following: infants affected by either congenital or chromosomal abnormalities or conditions that could interfere with growth, such as chronic lung disease (as defined based on the classification of Jobe and Bancalari), neurological disorders, metabolic, cardiac disease and abdominal surgery, renal failure and/or sepsis (defined as a positive blood culture).
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2015-01; Primary Completion 2017-02 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Protein balance | at hospital discharge (that is 35-36 post conceptional weeks)
  Protein balance will be determined according to nitrogen balance standard method and defined as the difference between daily nitrogen intake and daily urinary nitrogen excretion. Nitrogen intake will be measured from the amount of total protein intake (i.e. grams of nitrogen intake=grams of protein intake/6.25).
  Urinary urea nitrogen excretion will be considered representative of total nitrogen loss. Urinary urea will be calculated from urine specimens collected by cotton balls.

SECONDARY OUTCOMES:
Fat free mass content | Term corrected age (that is 40 post conceptional weeks)
  Body composition will be assessed by an air-displacement plethysmography system (PEA POD Infant Body Composition System, COSMED SRL, Roma, Italy). The PEA POD assesses fat mass and fat-free mass by direct measurements of body mass and volume and the application of a classic densitometric model.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Morlacchi, MD, Principal Investigator — Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico
Locations (1):
- NICU, Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico, Milan, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Morlacchi L, Roggero P, Gianni ML, Bracco B, Porri D, Battiato E, Menis C, Liotto N, Mallardi D, Mosca F. Protein use and weight-gain quality in very-low-birth-weight preterm infants fed human milk or formula. Am J Clin Nutr. 2018 Feb 1;107(2):195-200. doi: 10.1093/ajcn/nqx001. PMID 29529139